CLINICAL TRIAL: NCT06963138
Title: Comparative Study and Validation of New Methodologies for Measuring Addition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: WS10331; 2023-A00122-43 (Other: ANSM)
Record Dates: First submitted 2025-04-17; First posted 2025-05-08 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Presbyopia; Near Vision; Refraction Error
MeSH Terms: conditions — Presbyopia; Myopia; Refractive Errors | interventions — Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Validation of new addition measurement methodologies (Experimental)
  Interventions: Device: Visual Acuity; Device: Objective refraction; Device: Standard Subjective refraction; Device: Near vision examination and determination of additions; Device: Binocular vision tests; Device: Extended trial of addition

INTERVENTIONS:
Device: Visual Acuity — VA will be measured for near and distance vision with an Early Treatment Diabetic Retinopathy Study (ETDRS) chart
Device: Objective refraction — Objective refraction will be measured using an auto-kerato-refractometer/aberrometer
Device: Standard Subjective refraction — Standard subjective refraction for distance vision will be performed with Vision-R™
Device: Near vision examination and determination of additions — Near vision examination and determination of additions will be performed with Vision-R™. The following objective and subjective measurement methods will determine the values of the various additions:
  1. Determination of addition using the retinoscopy method (Add_OBJ)
  2. Randomization and administration of addition determination tests: FCC; R/G; PRA-NRA
Device: Binocular vision tests — The following measurements will be taken in trial glasses equipped with the final addition:
  1. Stereoscopic acuity measurement
  2. Measurement of the Near Point of Accommodation (PPA)
  3. Measurement of the Near Point of Convergence (PPC)
  4. Measurement of fusion reserves
  5. Measurement of prismatic rock
  6. Subjective questionnaire on the different methods used
Device: Extended trial of addition — The following measurements will be performed using trial glasses equipped with the final addition:
  1. Submission of the CISS questionnaire and distance adaptation
  2. Initial measurements of accommodative positioning and phorias
  3. Completion of three smartphone tasks: reading, memorization, and video viewing
  4. Final measurements of accommodative positioning and phorias
  5. Submission of the QoL questionnaire regarding visual discomfort during the trial.

SUMMARY:
The aim of this research is to collect comprehensive data on a presbyopic population that may require near vision correction, in order to identify the most useful tests to accurately determine the value of an addition.

DETAILED DESCRIPTION:
Refraction is the key point of an ophthalmic examination when visual correction is required for distance vision, as is determining the addition for near vision. These measurements can be obtained objectively and/or subjectively.

The addition for near vision is most often obtained using so-called subjective devices, i.e., by relying on the patient's responses.

The state of the accommodative system can, however, be measured objectively using instruments available to prescribers (retinoscopes, automatic refractometers, aberrometers, etc.). These measurements can be used in clinical practice as a solid basis for the initial assessment of the subject's refractive status during a comprehensive eye examination. However, these measurements are not sufficient to determine the optimal correction to prescribe for near vision, i.e., one that achieves sufficient visual acuity and comfort to ensure effectiveness for the tasks a person wishes to perform in their daily life.

Indeed, subjective tests are considered the gold standard for prescribers, particularly when it comes to near vision testing. Also, there are numerous procedures for determining the appropriate addition to prescribe, and a wide variety of practices is observed among prescribers around the world. It is often necessary to perform multiple tests to ensure the correct addition value to recommend.

The aim of this study is to find ways of approaching the value of the ideal addition as accurately as possible, based on several parameters: measurements representative of subjects' near vision habits, optometric measurements to determine near vision addition, and measurements related to binocular vision and symptomatology. This data collection will enable to identify the most effective combination of measurements in order to determine the optimal near vision addition for a subject.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer, fluent in French, willing to follow the protocol, able to read and understand the information form and give free and informed consent
* Aged 40 to 60 years
* Individual with monocular visual acuity ≥ +0.1 LogMAR with current corrections and pinhole if necessary
* Individual with a visual acuity difference ≤ 0.2 LogMAR with current corrections
* Individual with stable binocular vision in distance and near vision

Exclusion Criteria:

* Age < 40 years (i.e., no minors in accordance with Article L1121-7)
* Age > 60 years

All categories of people specifically protected under French law are excluded from this research (Articles L1121-5 to L1121-9 of the Public Health Code):

* Pregnant, childbearing, or breastfeeding women (Article L1121-5)
* Persons deprived of their liberty by a judicial or administrative decision and persons hospitalized without consent pursuant to Articles L. 3212-1 and L. 3213-1 who do not fall under the provisions of Article L. 1121-8 and persons admitted to a health or social care facility for purposes other than research
* Adults incapable or unable to express consent (Article L1121-8)
* Participants currently excluded from another study
* Participants unable to be contacted in case of emergency
* Person with strabismus
* Person with amblyopia
* Aphakic or pseudophakic person
* Person with vertical phoria > 1 PD
* Declared neurological deficit, including a history of epileptic disorders or sensory-motor coordination disorders, vestibular or cerebellar pathology (e.g., balance disorders)
* Declared severe ocular pathology, involving visual field loss, such as glaucoma, or involving loss of acuity and significant discomfort in dimly or excessively lit environments, such as retinitis pigmentosa, or declared and treated dry eye.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Subject's age | Day 1
  The subject's age is requested via the Case Report Form
Addition value given by the objective method | Day 1
  When you have presbyopia, the lens is no longer able to increase its power to accommodate near vision. It must then be helped by adding power for near vision, i.e., increasing the strength of the lens: this is called addition. The value of the addition is expressed in diopters (D) and is automatically measured by an auto-kerato-refractometer/aberrometer. It is an objective measure because it does not call upon the subject's responses when presented with acuity scales.
Addition value given by the subjective method | Day 1
  When you have presbyopia, the lens is no longer able to increase its power to accommodate near vision. It must then be helped by adding power for near vision, i.e., increasing the strength of the lens: this is called addition. The value of the addition is expressed in diopters (D) and is automatically measured by an autorefractometer. It is a subjective measure because it calls upon the subject's responses when presented with acuity scales.
Working distances for near vision | Day 1
  Several working distances are measured for near vision. The values of the distances are expressed in centimeters (cm).
  The various working distances for near vision are:
  * Harmon distance: the morphological distance from the elbow to the clenched fist
  * Revip distance (visuo-postural reflex): the subject is given a blank A4 sheet of paper and asked to hold it at their potential reading distance.
  * Desired distance: the distance at which a subject can read a Times 12 text on an A4 sheet of paper.

SECONDARY OUTCOMES:
Quality of Vision questionnaire (Qov) score | Day 1
  The QoV Questionnaire consists of a Rasch-tested, linear-scaled, 30-item instrument on three scales providing a QoV score in terms of symptom frequency, severity, and bothersome. It is suitable for measuring QoV in patients with all types of refractive correction, eye surgery, and eye disease that cause QoV problems.
  The QoV Questionnaire includes, 10 questions for each nature of evaluation (frequency, severity and bothersome) and 4 possible answers weighted by the values 0, 1, 2 or 3. The higher the score, the more frequently or intensely the symptom is perceived, or the more annoying it is, depending on the nature of the evaluation. Minimum score : 0 ; Maximum Score : 30.
CISS questionnaire (Convergence Insufficiency Symptom Survey) score | Day 1
  The CISS Questionnaire consists of a 14-item instrument providing a CISS score in terms of symptom frequency. Convergence Insufficiency is a condition in which a patient finds it difficult to maintain alignment of the eyes on a near object. The assessment of potential convergence difficulties in near vision may cause a person to look with just one eye at a time, or to see double.
  The Convergence Insufficiency Symptom Survey includes 5 questions relative to specific visual symptoms, with 5 possible answers weighted by the values 0, 1, 2, 3 or 4. The higher the score, the more frequently the symptom is perceived. Minimum Score : 0 ; Maximum Score : 60.

CONTACTS AND LOCATIONS:
Overall Officials: François Daniel, Principal Investigator — ESSILOR INTERNATIONAL - Division Instruments
Locations (1):
- Essilor International - Ci&T 2, Créteil, France